CLINICAL TRIAL: NCT05632003
Title: Uterocervical Angle Versus Cervical Length in The Prediction Of Spontaneous Preterm Birth In Women With History Of Spontaneous Preterm Birth A Prospective Observational Study
Brief Title: Uterocervical Angle in Prediction of Preterm Labor
Acronym: Preterm labor
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Elmaraghy, Lecturer, Ain Shams Maternity Hospital
Other Study IDs: 7
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preterm delivery occurs in about 5-18% of pregnancies before 37 weeks' gestation all over the world.It is associated with a high prevalence of neurological deficits, developmental disabilities and is a leading cause of infant and neonatal mortality.

Many of the methods used for predicting preterm birth has not been proven efficacy and is not currently recommended for use.The length of the cervix has been one of the most useful methods in predicting the risk of premature delivery. Detection rates may be improved if combined with other parameters such as the uterocervical angle as a new predictor of spontaneous preterm birth.

In this study we will compare between using the uterocervical angle and cervical length in the prediction of preterm labour.

DETAILED DESCRIPTION:
Preterm birth, defined as birth before 37 weeks of gestation, affects 5 to 18% of pregnancies. It is the leading cause of neonatal death and the second cause of childhood death below the age of 5 years. Preterm delivery (birth before 37 weeks' gestation) is further delineated into very early preterm (before 32 weeks), early preterm (32 0/7 to 33 6/7 weeks), and late preterm (34 0/7 to 36 6/7 weeks). It is logical to divide PTD into different subcategories: live-borns vs. intrauterine fetal deaths, singleton pregnancies vs. multiple pregnancies and spontaneous PTD vs. iatrogenic PTD. About 80% of all the preterm infants are live born singletons. The majority of these deliveries are spontaneous, due to onset of contractions or to spontaneously ruptured membranes. Conversely, iatrogenic preterm deliveries are due to the physician's decision to induce labor for maternal or fetal medical reasons. However, since the terminology varies, it is crucial to use clear definitions in all circumstances where the different phenotypical terms are used.

Preterm delivery is the consequence of four main mechanisms: activation of the maternal-fetal placental interaction with the hypothalamic-pituitary-adrenal axis, inflammation in the amniochorionic-decidual tissue, decidual hemorrhage and pathological distention of the myometrium. Although in most cases preterm births occur idiopathically, fetal, uterine, and placental factors as well as maternal chronic diseases, can affect preterm birth. It is estimated that of all cases of PTB, only 8.7% and 1.7- 2.3% of women, respectively, have the risk factors of prior PTB or significant cervical shortening in the midtrimester and would benefit from prophylactic therapy. A number of risk factors for preterm birth are known, but this does not mean that recognizing one of them in a pregnant woman before the 37th week means that a preterm birth will certainly begin. Knowledge of the risk factors allows for more intensive observation of the pregnant woman and gives obstetricians insight into what should be avoide . There are many maternal or fetal characteristics that have been associated with preterm birth, including maternal demographic characteristics, nutritional status, pregnancy history, present pregnancy characteristics, psychological characteristics, adverse behaviours, infection, uterine contractions and cervical length, and biological and genetic markers. Proposed techniques for detecting at-risk pregnancies include risk factor-based scoring systems, home uterine activity monitoring, maternal serum chemistries, salivary estriol, cervicovaginal chemistries, and amniotic fluid analytes. These modalities are characterized by either inadequate screening efficiencies, invasiveness, expense, or lack of commercial availability. Moreover, their use does not demonstrate reduced spontaneous preterm birth rates. Cervical length (CL) measured by transvaginal sonography (TVS) has been shown to be an effective predictor of spontaneous preterm birth (PTB). This finding has been confirmed in singleton and multiple gestations, in women with or without risk factors for preterm birth, and in asymptomatic women as well as women with preterm labor (PTL) or preterm prelabor rupture of the membranes (PPROM). The anterioruterocervical angle (aUCA) is a novel transvaginal ultrasonographic marker that showed evidence of being useful as a screening tool for spontaneous PTB. It can be used as an alternative to cervical length (CL) as screening method for sPTB. It involves measurement of the angle between the anterior lower uterine segment (LUS) and cervix. A wide, or obtuse, anterior uterocervical angle (aUCA) lends a more direct, linear outlet of uterine contents onto the cervix. A narrower, or acute, UCA supports an anatomical geometry that would exert less direct force on the internal os, which may be protective from cervical deformation. A wide aUCA ≥95ᶿ and ≥105ᶿ detected during the 2nd trimester was associated with an increased risk for sPTB<37 and <34 weeks, respectively. However, the studies that provided this evidence were retrospective and their results were heterogeneous. Our objective is to evaluate whether the anterior UCA can predict risk of sPTB in a general population of singletons and to evaluate its performance for predicting sPTB relative to CL.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy
2. History of spontaneous preterm birth
3. Recruitment at 16 to 24 weeks of pregnancy
4. Normal growth pattern evaluated by estimated fetal weight or abdominal circumference

Exclusion Criteria:

1. Medical disorders which can lead to uteroplacental insufficiency
2. Congenital uterine anomalies, as it may change the uterocervical angle.
3. Congenital fetal malformations detected on midtrimesteric anomaly scan
4. Pregnancy on IVF/ICSI
5. Smoking during pregnancy
6. History of cervical trauma
7. Preterm prelabor rupture of the membranes
8. Polyhydramnios
9. Cervical cerclage
10. Antepartum hemorrhage

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women attending the obstetrics outpatient clinic at AinShams university maternity hospital
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Early preterm birth | from 16 0/7 to 36 6/7 weeks of gestation
  birth between 32 0/7 and 33 6/7 weeks of gestation

SECONDARY OUTCOMES:
Late preterm birth | from 16 0/7 to 36 6/7 weeks of gestation
  birth between 34 0/7 and 36 6/7 weeks of gestation

OTHER OUTCOMES:
Very early preterm birth | from 16 0/7 to 36 6/7 weeks of gestation
  birth before 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S Elsokkary, MD, Study Director — Ainshams university maternity hospital
Locations (1):
- AinShams university maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berghella V, Palacio M, Ness A, Alfirevic Z, Nicolaides KH, Saccone G. Cervical length screening for prevention of preterm birth in singleton pregnancy with threatened preterm labor: systematic review and meta-analysis of randomized controlled trials using individual patient-level data. Ultrasound Obstet Gynecol. 2017 Mar;49(3):322-329. doi: 10.1002/uog.17388. Epub 2017 Feb 8. PMID 27997053
- [Background] DeFranco EA, Lewis DF, Odibo AO. Improving the screening accuracy for preterm labor: is the combination of fetal fibronectin and cervical length in symptomatic patients a useful predictor of preterm birth? A systematic review. Am J Obstet Gynecol. 2013 Mar;208(3):233.e1-6. doi: 10.1016/j.ajog.2012.12.015. Epub 2012 Dec 12. PMID 23246314
- [Background] Di Renzo GC, Cabero Roura L, Facchinetti F, Helmer H, Hubinont C, Jacobsson B, Jorgensen JS, Lamont RF, Mikhailov A, Papantoniou N, Radzinsky V, Shennan A, Ville Y, Wielgos M, Visser GHA. Preterm Labor and Birth Management: Recommendations from the European Association of Perinatal Medicine. J Matern Fetal Neonatal Med. 2017 Sep;30(17):2011-2030. doi: 10.1080/14767058.2017.1323860. No abstract available. PMID 28482713
- [Background] Dziadosz M, Bennett TA, Dolin C, West Honart A, Pham A, Lee SS, Pivo S, Roman AS. Uterocervical angle: a novel ultrasound screening tool to predict spontaneous preterm birth. Am J Obstet Gynecol. 2016 Sep;215(3):376.e1-7. doi: 10.1016/j.ajog.2016.03.033. Epub 2016 Mar 24. PMID 27018466
- [Background] Farras Llobet A, Higueras T, Calero IZ, Regincos Marti L, Maiz N, Goya MM, Carreras E. Prospective evaluation of the uterocervical angle as a predictor of spontaneous preterm birth. Acta Obstet Gynecol Scand. 2020 Nov;99(11):1511-1518. doi: 10.1111/aogs.13879. Epub 2020 Jun 3. PMID 32311754
- [Background] Halimi Asl AA, Safari S, Parvareshi Hamrah M. Epidemiology and Related Risk Factors of Preterm Labor as an obstetrics emergency. Emerg (Tehran). 2017;5(1):e3. Epub 2017 Jan 8. PMID 28286810
- [Background] Kagan KO, Sonek J. How to measure cervical length. Ultrasound Obstet Gynecol. 2015 Mar;45(3):358-62. doi: 10.1002/uog.14742. Epub 2015 Jan 29. No abstract available. PMID 25632014
- [Background] Khamees RE, Khattab BM, Elshahat AM, Taha OT, Aboelroose AA. Uterocervical angle versus cervical length in the prediction of spontaneous preterm birth in singleton pregnancy. Int J Gynaecol Obstet. 2022 Feb;156(2):304-308. doi: 10.1002/ijgo.13629. Epub 2021 Feb 23. PMID 33507541
- [Background] Pawelec M, Palczynski B, Krzemieniewska J, Karmowski M, Korys J, Latkowski K, Karmowski A. Initiation of preterm labor. Adv Clin Exp Med. 2013 Mar-Apr;22(2):283-8. PMID 23709385
- [Background] Romero R, Dey SK, Fisher SJ. Preterm labor: one syndrome, many causes. Science. 2014 Aug 15;345(6198):760-5. doi: 10.1126/science.1251816. Epub 2014 Aug 14. PMID 25124429
- [Background] Rundell K, Panchal B. Preterm Labor: Prevention and Management. Am Fam Physician. 2017 Mar 15;95(6):366-372. PMID 28318214
- [Background] Sen C. Preterm labor and preterm birth. J Perinat Med. 2017 Nov 27;45(8):911-913. doi: 10.1515/jpm-2017-0298. No abstract available. PMID 29055176
- [Background] Wax JR, Cartin A, Pinette MG. Biophysical and Biochemical Screening for the Risk of Preterm Labor: An Update. Clin Lab Med. 2016 Jun;36(2):369-83. doi: 10.1016/j.cll.2016.01.019. Epub 2016 Mar 25. PMID 27235918
- [Derived] Elmaraghy AM, Shaaban SMA, Elsokkary MS, Elshazly ISMA. Uterocervical angle versus cervical length in the prediction of spontaneous preterm birth in women with history of spontaneous preterm birth: a prospective observational study. BMC Pregnancy Childbirth. 2023 Sep 13;23(1):658. doi: 10.1186/s12884-023-05977-9. PMID 37704977